CLINICAL TRIAL: NCT00161005
Title: Benefits and Costs in Two Different Strategies for Treating Acute Myocardial Infarction With ST-Elevation.
Brief Title: Norwegian Study on District Treatment of ST-Elevation Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Helse Innlandet (Unknown)
Responsible Party: dr.Sigrun Halvorsen, Hjertemed avd., UUH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2935-0304 (UUS); 2004-162 (Helse Oest)
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2009-04-17 (Estimated); Status verified 2009-04

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; Fibrinolysis; Health effects /Quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: PCI — Immediate transport to invasive center after thrombolysis

SUMMARY:
In the district areas of Norway patients with acute myocardial infarction with ST-elevation, are treated with thrombolysis. An increasing part of them receives thrombolysis before arrival to the local hospital.Usually these patients have been sent to an invasive center if thrombolysis fails or the patient gets ischemic symptoms during the stay.

This study will compare this strategy against immediate transportation to an invasive center after the patient has received thrombolysis.

ELIGIBILITY:
Inclusion Criteria:

* Duration of painless than 6 hours.
* ST-segment elevation of at least 0.1 mV in two or more extremity leads or at least 0.2 mV in two or more precordial leads.
* The patient is getting thrombolysis.
* Time to reach an invasive center is more than 1 hour.
* Age 18-75 years.

Exclusion Criteria:

* Known serious renal failure (creatinin > 250 mmol/l)
* Pregnancy
* Cardiogenic chock
* Life threatening arrythmias
* Other serious diseases with life expectancy less than 1 year.
* Inability to perform an informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2005-02; Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Death , myocardial infarction ,stroke or ischemia during 12 months. | 12 months
Costs during 12 months. | 12 months

SECONDARY OUTCOMES:
Size of infarction. | 3 months
Complications | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Sigrun Halvorsen@uus.no, dr.med, Principal Investigator — UUS, Oslo, Norway
Locations (1):
- Ulleval University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Bohmer E, Kristiansen IS, Arnesen H, Halvorsen S. Health-related quality of life after myocardial infarction, does choice of method make a difference? Scand Cardiovasc J. 2014 Aug;48(4):216-22. doi: 10.3109/14017431.2014.923581. Epub 2014 Jun 26. PMID 24828790
- [Derived] Halvorsen S, Seljeflot I, Weiss T, Bohmer E, Arnesen H. Inflammatory and thrombotic markers in patients with ST-elevation myocardial infarction treated with thrombolysis and early PCI: a NORDISTEMI substudy. Thromb Res. 2012 Sep;130(3):495-500. doi: 10.1016/j.thromres.2012.04.016. Epub 2012 May 17. PMID 22607887
- [Derived] Bohmer E, Kristiansen IS, Arnesen H, Halvorsen S. Health and cost consequences of early versus late invasive strategy after thrombolysis for acute myocardial infarction. Eur J Cardiovasc Prev Rehabil. 2011 Oct;18(5):717-23. doi: 10.1177/1741826711398425. Epub 2011 Feb 18. PMID 21450598
- [Derived] Mistry N, Bohmer E, Hoffmann P, Muller C, Bjornerheim R, Kjeldsen SE, Halvorsen S. Left ventricular function in acute myocardial infarction treated with thrombolysis followed by early versus late invasive strategy. Am Heart J. 2010 Jul;160(1):73-9. doi: 10.1016/j.ahj.2010.04.011. PMID 20598975
- [Derived] Bohmer E, Hoffmann P, Abdelnoor M, Arnesen H, Halvorsen S. Efficacy and safety of immediate angioplasty versus ischemia-guided management after thrombolysis in acute myocardial infarction in areas with very long transfer distances results of the NORDISTEMI (NORwegian study on DIstrict treatment of ST-elevation myocardial infarction). J Am Coll Cardiol. 2010 Jan 12;55(2):102-10. doi: 10.1016/j.jacc.2009.08.007. Epub 2009 Sep 10. PMID 19747792
- [Derived] Bohmer E, Arnesen H, Abdelnoor M, Mangschau A, Hoffmann P, Halvorsen S. The NORwegian study on DIstrict treatment of ST-elevation myocardial infarction (NORDISTEMI). Scand Cardiovasc J. 2007 Jan;41(1):32-8. doi: 10.1080/14017430601153472. PMID 17365975